CLINICAL TRIAL: NCT04143256
Title: An Open-Label, Multi-Center Study to Evaluate Selected Constituents in the Exhaled Breath Samples From the Use of JUUL Nicotine Salt Pod System Product (5% and 3% Virginia Tobacco, Mint, Mango, Menthol) Users and Conventional Cigarettes (Non-Menthol and Menthol Flavors)
Brief Title: Evaluating Selected Constituents in the Exhaled Breath Samples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juul Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PROT-00109
Record Dates: First submitted 2019-10-24; First posted 2019-10-29 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Electronic Cigarette Use; Cigarette Use, Electronic; Tobacco Use; Tobacco Smoking
Keywords: Electronic Nicotine Delivery; Combustible Cigarettes; Nicotine; Exhaled Breath
MeSH Terms: conditions — Vaping; Tobacco Use; Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: Four crossover groups and two single arm groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group I (Experimental): Subjects with ENDS user history may be randomized to use JUUL ENDS 5% Virginia Tobacco and 3% Virginia Tobacco
  Interventions: Other: JUUL ENDS 5% Virginia Tobacco; Other: JUUL 3% Virginia Tobacco ENDS
- Group II (Experimental): Subjects with ENDS user history may be randomized to use JUUL ENDS 5% Mint and 3% Mint
  Interventions: Other: JUUL 5% Mint ENDS; Other: JUUL 3% Mint ENDS
- Group III (Experimental): Subjects with ENDS user history may be randomized to use JUUL ENDS 5% Menthol and 3% Menthol
  Interventions: Other: JUUL 5% Menthol ENDS; Other: JUUL 3% Menthol ENDS
- Group IV (Experimental): Subjects with ENDS user history may be randomized to use JUUL ENDS 5% Mango and 3% Mango
  Interventions: Other: JUUL 5% Mango ENDS; Other: JUUL 3% Mango ENDS
- Group V (Experimental): Subjects with cigarette user history will be assigned to use US Cigarette, Non-Menthol Flavor (Marlboro Gold King Size)
  Interventions: Other: US Cigarette, Non-menthol - Marlboro Gold King Size
- Group VI (Experimental): Subjects with cigarette user history will be assigned to use US Cigarette, Menthol Flavor (Newport King Size)
  Interventions: Other: US Cigarette, Menthol - Newport King Size

INTERVENTIONS:
Other: JUUL ENDS 5% Virginia Tobacco — JUUL ENDS Virginia Tobacco 5% nicotine strength
  Arms: Group I
Other: JUUL 3% Virginia Tobacco ENDS — JUUL ENDS Virginia Tobacco 3% nicotine strength
  Arms: Group I
Other: JUUL 5% Mint ENDS — JUUL ENDS Mint 5% nicotine strength
  Arms: Group II
Other: JUUL 3% Mint ENDS — JUUL ENDS Mint 3% nicotine strength
  Arms: Group II
Other: JUUL 5% Menthol ENDS — JUUL ENDS Menthol 5% nicotine strength
  Arms: Group III
Other: JUUL 3% Menthol ENDS — JUUL ENDS Menthol 3% nicotine strength
  Arms: Group III
Other: JUUL 5% Mango ENDS — JUUL ENDS Mango 5% nicotine strength
  Arms: Group IV
Other: JUUL 3% Mango ENDS — JUUL ENDS Mango 3% nicotine strength
  Arms: Group IV
Other: US Cigarette, Non-menthol - Marlboro Gold King Size — US Cigarette, Non-menthol - Marlboro Gold King Size
  Arms: Group V
Other: US Cigarette, Menthol - Newport King Size — US Cigarette, Menthol - Newport King Size
  Arms: Group VI

SUMMARY:
An Open-Label, Multi-Center Study to Evaluate Selected Constituents in the Exhaled Breath Samples From the Use of JUUL Nicotine Salt Pod System Product (5% and 3% Virginia Tobacco, Mint, Mango, Menthol) Users and Conventional Cigarettes (Non-Menthol and Menthol Flavors)

DETAILED DESCRIPTION:
The objective of this study is to evaluate the baseline-adjusted level of selected constituents in the exhaled breath sample (EBS) between the two JUUL NSPS products (5% vs 3% nicotine by weight) for Virginia Tobacco, Mint, Mango and Menthol flavor and to compare the change in absolute level of selected constituents in EBS before and after the use of JUUL NSPS (5% and 3% nicotine by weight; Virginia Tobacco, Mint, Mango, Menthol flavors) to the change in absolute level of selected constituents before and after the use of menthol and non-menthol cigarettes.

Subjects will be screened for participation in the trial up to 28 days before Day 1. Along with screening procedures, all subjects will receive training on EBS collection procedures. All subjects will be further trained on the CPS using a training video and site instructions. Trained subjects will have the opportunity to try the JUUL NSPS.

Eligible subjects will be scheduled for a Day 1 clinic visit. Within 24 to 48 hours prior to Check-in, the clinic staff will provide a courtesy phone call to subjects to remind them to abstain from the use of alcohol, any nicotine-containing products and mint/mentholated products for at least 12 hours prior and xanthines/caffeine for at least 24 hours prior to screening and Day 1.

Following completion of the check-in events, including re-instruction on the EBS sample collection technique and CPS instructions, subjects will participate in the exhaled breath collection test sessions.

Groups I - IV will complete two periods of baseline and test sample collections with a 3-hour break in between each period. Each period will consist of two baseline samples (the first for analysis of nicotine, propylene glycol and glycerin and the second for analysis of acetaldehyde, acrolein, benzoic acid, formaldehyde, and menthol), followed by product use, and then two test samples (similar to baseline). Exhaled CO will be measured before the first baseline sample, after the second baseline sample, before the first test sample and after the second test sample. Pods used during the test sessions will be weighed before and after use.

Groups V and VI will complete only one period of baseline and test sample collections, consisting of two baseline sample collections and two test sample collections similar to that noted above.

A follow-up phone call with subjects will be made the day after Check-out (or early withdrawal). Provided there are no adverse events which require further attention, the subject's participation in the trial will be complete.

ELIGIBILITY:
Inclusion Criteria:

1. Be a healthy male or female aged 21 - 65 years, inclusive, at the time of signing the informed consent.
2. Be informed of the nature of the study, agree to and are able to read, review, and sign the informed consent document prior to any study procedures. The informed consent document will only be available in English. Therefore, the volunteer must have the ability to read and communicate in English in order to participate in the study.
3. Complete the screening process up to 28 days prior to Day 1.
4. Satisfy the user definitions of either cigarette user or ENDS/closed system user.
5. Agree to abide by the study restrictions.
6. Agree to abstain from use of alcohol 12 hours before the start of Day 1 for Groups I through VI.
7. Agree to abstain from use of any nicotine products 12 hours before the start of study day 1 for Groups I through VI.
8. Agree to not consume any mint or menthol flavor products (e.g., chewing gum, mouth wash, toothpaste, etc.) 12 hours before the start of testing for Groups I through VI.
9. Have a positive urine cotinine result at screening of >200 ng/ml.
10. A female subject of childbearing potential must have been using one (1) of the following forms of contraception and agree to continue using it through completion of the trial:

    * hormonal (e.g., oral, vaginal ring, transdermal patch, implant, or injection) consistently for at least 3 months prior to Day 1;
    * double barrier method (e.g., condom with spermicide, diaphragm with spermicide) at screening.
    * intrauterine device for at least 3 months prior to Day 1;
    * a partner who has been vasectomized for at least 6 months prior to Day 1;
    * abstinence beginning at least 6 months prior to screening.
11. A female subject of non childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to Day 1:

    * hysteroscopic sterilization;
    * bilateral tubal ligation or bilateral salpingectomy;
    * hysterectomy;
    * bilateral oophorectomy;
    * Or be postmenopausal with amenorrhea for at least 1 year prior to Day 1.
12. Be judged by the Investigator to be in good general health as documented by the medical history, physical examination (including but may not be limited to an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems), vital sign assessments and by general observations. Any abnormalities or deviations outside the normal ranges for any clinical testing (e.g. vital signs) can be repeated at the discretion of the Investigator and judged to be not clinically significant for study participation.

Exclusion Criteria:

1. Report receiving any investigational product, participated in any previous clinical study for an investigational drug, device, biologic, or tobacco product within 30 days prior to screening.
2. Report at screening using both ENDS and conventional cigarettes (menthol or non-menthol) (dual users), or use of other inhaled products (such as, but not limited to cannabis) in the past 3 months.
3. For ENDS users, be unable to perform CPS or incapable of drawing down the pod weight by 20-60mg after 3 attempts at screening.
4. If female, be pregnant, have a positive urine pregnancy test at screening, be lactating, breast feeding, or intend to become pregnant during the time period from screening through the end of the study.
5. Have any clinically significant results from physical examinations and vital signs assessments, as judged by the Investigator.
6. Have a systolic blood pressure < 90 mmHg or > 150 mmHg, diastolic blood pressure < 40 mmHg or > 95 mmHg, or heart rate < 40 bpm or > 99 bpm at screening.
7. Report a clinically significant illness during the 30 days prior to enrollment, as determined by the Investigator.
8. Report a history of drug or alcohol addiction or abuse within the past 1 year.
9. Have a positive screen for alcohol or drugs of abuse at screening or at check-in on Day 1.
10. Have a body mass index (BMI) greater than 40 kg/m2 or less than 18 kg/m2 at screening.
11. Have used prescription anti-diabetic medication and/or insulin therapy within 12 months of screening.
12. Have taken medication for depression, asthma, or chronic obstructive pulmonary disease within 6 months of screening.
13. Have used prescription or over-the-counter bronchodilator medication (e.g., inhaled or oral β-agonists) within 6 months of screening.
14. Be breast-feeding or pregnant female subjects (confirmed by a positive pregnancy test). Female subjects, who are considered women of child bearing potential (WOCBP) and sexually active, must be willing and able to use an acceptable method of contraception from screening through the end of the study.
15. Have experienced an allergic reaction following previous e-cigarette use or with exposure to any primary components of the e-liquids (nicotine, flavor, benzoic acid, propylene glycol, and/or glycerol.
16. Be or have a first-degree relative (i.e. parent, sibling or child) who is a current employee of CRO, Sponsor, or site.
17. In the opinion of an Investigator, be deemed not eligible to participate in this study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Evaluate Absolute Change from Baseline Level | Up to 6-hours
  The absolute change from baseline level of nicotine for each subject.
Evaluate Absolute Change from Baseline Level | Up to 6-hours
  The absolute change from baseline level of propylene glycol for each subject.
Evaluate Absolute Change from Baseline Level | Up to 6-hours
  The absolute change from baseline level of vegetable glycerin for each subject.
Evaluate Absolute Change from Baseline Level | Up to 6-hours
  The absolute change from baseline level of acetaldehyde for each subject.
Evaluate Absolute Change from Baseline Level | Up to 6-hours
  The absolute change from baseline level of acrolein for each subject.
Evaluate Absolute Change from Baseline Level | Up to 6-hours
  The absolute change from baseline level of benzoic acid for each subject.
Evaluate Absolute Change from Baseline Level | Up to 6-hours
  The absolute change from baseline level of formaldehyde for each subject.
Evaluate Absolute Change from Baseline Level | Up to 6-hours
  The absolute change from baseline level of menthol for each subject.
Evaluate Absolute Change from Baseline Level | Up to 6-hours
  The absolute change from baseline level of carbon monoxide for each subject.

SECONDARY OUTCOMES:
Compare the change between baseline and post-baseline levels | Up to 6-hours
  Compare the change between baseline and post-baseline levels of nicotine for each subject.
Compare the change between baseline and post-baseline levels | Up to 6-hours
  Compare the change between baseline and post-baseline levels of propylene glycol for each subject.
Compare the change between baseline and post-baseline levels | Up to 6-hours
  Compare the change between baseline and post-baseline levels of vegetable glycerin for each subject.
Compare the change between baseline and post-baseline levels | Up to 6-hours
  Compare the change between baseline and post-baseline levels of acetaldehyde for each subject.
Compare the change between baseline and post-baseline levels | Up to 6-hours
  Compare the change between baseline and post-baseline levels of acrolein for each subject.
Compare the change between baseline and post-baseline levels | Up to 6-hours
  Compare the change between baseline and post-baseline levels of benzoic acid for each subject.
Compare the change between baseline and post-baseline levels | Up to 6-hours
  Compare the change between baseline and post-baseline levels of formaldehyde for each subject.
Compare the change between baseline and post-baseline levels | Up to 6-hours
  Compare the change between baseline and post-baseline levels of menthol for each subject.
Compare the change between baseline and post-baseline levels | Up to 6-hours
  Compare the change between baseline and post-baseline levels of carbon monoxide for each subject.
Change in weight | Up to 45
  Change in the weight of JUUL pods before and after the usage.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Frontage Clinical Services, Secaucus, New Jersey
  - Rose Research Center, Charlotte, North Carolina
  - Rose Research Center, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD to other researchers.

REFERENCES:
- [Derived] Oldham MJ, Bailey PC, Castro N, Lang Q, Salehi A, Rostami AA. Prediction of potential passive exposure from commercial electronic nicotine delivery systems using exhaled breath analysis and computational fluid dynamic techniques. J Breath Res. 2021 Oct 5;15(4). doi: 10.1088/1752-7163/ac2884. PMID 34544050